CLINICAL TRIAL: NCT04257929
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 2 Study to Evaluate the Safety and Efficacy of Pitolisant in Patients With Prader-Willi Syndrome, Followed by an Open Label Extension
Brief Title: A Phase 2 Study to Evaluate the Safety and Efficacy of Pitolisant in Patients With Prader-Willi Syndrome, Followed by an Open Label Extension
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Harmony Biosciences Management, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HBS-101-CL-002
Record Dates: First submitted 2020-01-29; First posted 2020-02-06 (Actual); Results first posted 2025-10-22 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Prader-Willi Syndrome
Keywords: PWS
MeSH Terms: conditions — Prader-Willi Syndrome | interventions — pitolisant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Double-Blind Treatment Phase Lower Dose Pitolisant (Active Comparator): Pediatric patients (6 to less than 12 years of age):
  Week 1: 4.45 mg pitolisant administered once daily in the morning; Week 2: 8.9 mg pitolisant administered once daily in the morning; Weeks 3 through 11: 8.9 mg pitolisant administered once daily in the morning.
  Adolescent patients (12 to less than 18 years of age):
  Week 1: 4.45 mg pitolisant administered once daily in the morning; Week 2: 8.9 mg pitolisant administered once daily in the morning; Weeks 3 through 11: 13.35 mg pitolisant administered once daily in the morning.
  Adult patients (18 to 65 years of age):
  Week 1: 4.45 mg pitolisant administered once daily in the morning; Week 2: 8.9 mg pitolisant administered once daily in the morning; Weeks 3 through 11: 17.8 mg pitolisant administered once daily in the morning.
  Interventions: Drug: Pitolisant oral tablets
- Double-Blind Treatment Phase Higher Dose Pitolisant (Active Comparator): Pediatric patients (6 to less than 12 years of age):
  Week 1: 4.45 mg pitolisant administered once daily in the morning; Week 2: 8.9 mg pitolisant administered once daily in the morning; Weeks 3 through 11: 17.8 mg pitolisant administered once daily in the morning.
  Adolescent patients (12 to less than 18 years of age):
  Week 1: 8.9 mg pitolisant administered once daily in the morning; Week 2: 17.8 mg pitolisant administered once daily in the morning; Weeks 3 through 11: 26.7 mg pitolisant administered once daily in the morning.
  Adult patients (18 to 65 years of age):
  Week 1: 8.9 mg pitolisant administered once daily in the morning; Week 2: 17.8 mg pitolisant administered once daily in the morning; Weeks 3 through 11: 35.6 mg pitolisant administered once daily in the morning.
  Interventions: Drug: Pitolisant oral tablets
- Double-Blind Treatment Phase Placebo (Placebo Comparator): Pediatric patients (6 to less than 12 years of age):
  Week 1: Matching placebo tablets; Week 2: Matching placebo tablets; Weeks 3 through 11: Matching placebo tablets
  Adolescent patients (12 to less than 18 years of age):
  Week 1: Matching placebo tablets; Week 2: Matching placebo tablets; Weeks 3 through 11: Matching placebo tablets
  Adult patients (18 to 65 years of age):
  Week 1: Matching placebo tablets; Week 2: Matching placebo tablets; Weeks 3 through 11: Matching placebo tablets
  Interventions: Drug: Placebo oral tablet
- Open-Label Pitolisant (Other): Age-based dosing (prior to implementation of amendment 6) or weight-based dosing (after implementation of amendment 6)
  Interventions: Drug: Pitolisant oral tablets

INTERVENTIONS:
Drug: Pitolisant oral tablets — Pitolisant 4.45 mg or 17.8 mg tablets
  Arms: Double-Blind Treatment Phase Higher Dose Pitolisant; Double-Blind Treatment Phase Lower Dose Pitolisant; Open-Label Pitolisant
Drug: Placebo oral tablet — Matching placebo tablets
  Arms: Double-Blind Treatment Phase Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety and efficacy of pitolisant compared with placebo in treating excessive daytime sleepiness (EDS) in patients with Prader Willi syndrome (PWS) ages 6 to 65 years.

DETAILED DESCRIPTION:
The study will consist of a Screening Period, an 11-week Double-Blind Treatment Phase (including a 3-week Titration Period and an 8-week Stable Dose Period), and an optional Open Label Extension (OLE) Phase. The OLE Phase will be multi-year in duration and will continue until the Sponsor elects to terminate the study.

Approximately 60 patients ages 6 to 65 years who meet all eligibility criteria will be randomized at the Baseline Visit in a 1:1:1 ratio to lower dose pitolisant, higher dose pitolisant, or matching placebo. In the Double-Blind Treatment Phase, patients will be titrated to their randomized stable dose of study drug during the 3-week Titration Period.

After completion of the 3-week Titration Period, patients will continue to take study drug at their randomized stable dose once daily in the morning upon wakening for an additional 8 weeks of blinded treatment (Stable Dose Period). The duration of the Double-Blind Treatment Phase will be 11 weeks.

Following the 11-week Double-Blind Treatment Phase, eligible patients will be given the opportunity to participate in an optional OLE Phase. During the OLE Phase, all eligible patients will receive treatment with open-label pitolisant and will undergo titration during a 3-week Titration Period to a maximum target dose as specified in the protocol. At the end of the 3-week Titration Period, patients will continue to take their target dose of pitolisant once daily in the morning upon wakening until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Is able to provide voluntary, written informed consent (patient or parent[s]/legal guardian[s]) and, where applicable, voluntary, written assent (patient, as appropriate).
2. Has a diagnosis of PWS confirmed by genetic testing and/or patient medical records. Genetic testing will be provided by the Sponsor, if not confirmed based on the review of the patient's medical records.
3. Male or female patients ages 6 to 65 years at the time of enrollment.
4. Demonstrates adequate sleep duration via patient sleep diary during Screening, defined as at least 8 hours of sleep per night for patients ages 6 to <12 years, at least 7 hours for patients ages 12 to <18 years, or at least 6 hours for patients ages ≥18 years, based on the mean number of hours from up to 14 nights (at least 7 nights must be recorded for evaluation).
5. Has EDS as determined by Epworth Sleepiness Scale for Children and Adolescents (ESS-CHAD) (parent/caregiver version) score of ≥12.
6. If taking hormone treatments (including growth hormone, testosterone, and estrogen supplements) and/or allowed chronic concomitant medication or supplements, patient must be on a stable dose of these medications for 3 months prior to randomization and for the duration of the Double-Blind Treatment Phase of the study; a 10% variability in hormone dose is allowed.
7. If taking a wake-promoting treatment that could affect EDS (including stimulants, modafinil, and armodafinil), must be on a stable dose for at least 28 days prior to Screening and remain on a stable dose during the Double-Blind Treatment Phase of the study (dose adjustments will be permitted in the OLE Phase) or agree to wash out of treatment for 5 half-lives or 14 days, whichever is longer.
8. If taking a chronically administered sedating medication for management of behavioral manifestations (e.g., hypnotics, benzodiazepines, antipsychotics, alpha agonists, anticholinergics, and antidepressants) must be on a stable dose for at least 28 days prior to Screening and remain on a stable dose during the Double-Blind Treatment Phase of the study (dose adjustments will be permitted in the OLE Phase) or agree to wash out of treatment for 5 half-lives or 14 days, whichever is longer.
9. If using cannabidiol and/or tetrahydrocannabinol, patient must be on a stable dose for 28 days prior to randomization and agree to continue the stable dose for the duration of the Double-Blind Treatment Phase of the study (dose adjustments will be permitted in the OLE Phase).
10. If taking oxytocin or carbetocin, patient must be on a stable dose during the 28 days prior to randomization and agree to continue the stable dose for the duration of the Double-Blind Treatment Phase of the study (dose adjustments will be permitted in the OLE Phase) or agree to wash out of treatment for 5 half-lives or 14 days, whichever is longer.
11. A patient who is a female of child-bearing potential (FCBP) must have a negative serum pregnancy test at the Screening Visit and a negative urine pregnancy test at the Baseline Visit and agree to remain abstinent or use an effective method of nonhormonal contraception to prevent pregnancy for the duration of the study and for 21 days after final dose of study drug.
12. Has a consistent caregiver (preferably the same person throughout the Double-Blind Treatment Phase of the study) who is willing and able to complete the required assessments.
13. In the opinion of the Investigator, patient/parent(s)/legal guardian(s) is capable of understanding and complying with the requirements of the protocol and administration of oral study drug.

Exclusion Criteria:

1. Has a diagnosis of another genetic or chromosomal disorder distinct from PWS.
2. Has untreated obstructive sleep apnea (OSA) or is at high risk for OSA based on medical history and clinical assessment; or, has another relevant underlying sleep disorder that in the opinion of the Investigator is the primary contributing factor to the patient's EDS.
3. Consistently consumes >600 mg of caffeine per day and is unable/unwilling to reduce caffeine intake to <600 mg per day for the duration of the Double-Blind Treatment Phase of the study; caffeine intake should remain consistent during Screening and throughout the Double-Blind Treatment Phase of the study.
4. Does not agree to discontinue any prohibited medication or substance listed in the protocol.
5. Participation in an interventional research study involving another investigational medication or device in the 28 days prior to enrollment and for the duration of the Double-Blind Treatment Phase of the study, unless the Investigator consults with the Medical Monitor and obtains written approval for the patient to enroll; patients who complete a washout of an investigational medication of at least 5 half-lives or 14 days (whichever is longer) may be enrolled in the Double-Blind Treatment Phase of the study. Patients considering participation in another interventional research study in the OLE Phase must consult with the Investigator who will consult with the Medical Monitor.
6. Has a primary psychiatric diagnosis with current active symptoms of psychosis or schizophrenia.
7. Has a diagnosis of end-stage renal disease (estimated glomerular filtration rate [eGFR] of <15 mL/minute/1.73 m²) or severe hepatic impairment (Child-Pugh C).
8. Has a diagnosis of moderate or severe renal impairment (eGFR ≥15 to ≤59 mL/minute/1.73 m²) or moderate hepatic impairment (Child-Pugh B) at Screening or during the Double-Blind Treatment Phase.
9. Has abnormal laboratory values at Screening that are clinically significant as determined by the Investigator.
10. Has a known history of long QT syndrome or any significant history of a serious abnormality of the electrocardiogram (ECG; e.g., recent myocardial infarction, clinically significant arrhythmia) or QT interval corrected for heart rate according to Fridericia's formula (QTcF) >442 ms for patients ages 0 to <10 years and >439 ms for patients ages 10 to <20 years, regardless of gender, and >450 ms for male patients and >470 ms for female patients ages 20 to 65 years. (ECG QTcF = QT/3√ RR) (Mason et al 2007).
11. Has a family history of sudden/unexplained death, cardiac death, or death from a primary dysrhythmia potentially associated with QT prolongation in any family member.
12. If receiving any new or initiating a change in allied health therapies or interventions for symptoms of PWS, must be on a stable course of therapy for at least 28 days prior to randomization.
13. Has a current or recent (within one year) history of a substance use disorder or dependence disorder, including alcohol and caffeine use disorders as defined in the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-V).
14. Has planned surgery during the Double-Blind Treatment Phase of the study; planned surgery is permitted during the OLE Phase.
15. Is receiving a concomitant medication that is known to be a strong cytochrome P450 (CYP) 2D6 inhibitor, a strong CYP3A4 inducer, or a centrally acting histamine 1 (H1) receptor antagonist; patients who complete a washout of these medications of at least 5 half-lives or 14 days (whichever is longer) can be enrolled in the Double-Blind Treatment Phase of the study. Use of strong CYP2D6 inhibitors and strong CYP3A4 inducers is allowed during the OLE Phase; however, adjustment of pitolisant dose is required. Although not prohibited during the OLE Phase of the study, use of H1 receptor antagonists should be avoided.
16. Is receiving a medication known to prolong the QT interval.
17. Has a significant risk of committing suicide based on history, routine psychiatric examination, Investigator's judgment, or an answer of "yes" on any question other than questions 1 to 3 on the Very Young Child/Cognitively Impaired-Lifetime Recent Columbia-Suicide Severity Rating Scale (C SSRS).
18. Has a history of seizures that have recently (within 6 months) been treated with antiepileptic medications that are strong CYP3A4 inducers. Patients with a history of seizures must have a stable seizure history (e.g., frequency and severity) for at least 6 months prior to enrollment.
19. Is currently breastfeeding or planning to breastfeed over the course of the study. Lactating women must agree not to breastfeed for the duration of the study (Double-Blind Treatment Phase and OLE Phase) and for 21 days after final dose of study drug.
20. Based on the judgment of the Investigator, patient is unsuitable for the study for any reason, including but not limited to unstable or uncontrolled medical conditions (including psychiatric and neurological conditions) or a medical condition that might interfere with the conduct of the study, confound interpretation of study results, pose a health risk to the patient, or compromise the integrity of the study.

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2028-09-07 (Estimated)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Rady Children's Hospital - San Diego, San Diego, California
  - Sleep Medicine Specialists of California, San Ramon, California
  - Santa Monica Clinical Trials, Santa Monica, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours Alfred I duPont Hospital for Children, Wilmington, Delaware
  - University of Florida College of Medicine, Gainesville, Florida
  - Ann and Robert H Lurie Children's Hospital, Chicago, Illinois
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CTI, Cincinnati, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Children's Hospital/Baylor College of Medicine, Houston, Texas
  - Road Runner Research, San Antonio, Texas

REFERENCES:
- [Derived] Revana A, Bhattacharjee R, Miller JL, Chidekel A, Khanna P, Ratnam S, Runyan G, Bauer E, Davis Rapchak K, Seiden D, Budur K, Dayno JM. A proof-of-concept study of pitolisant for excessive daytime sleepiness in patients with Prader-Willi syndrome. J Clin Sleep Med. 2025 Nov 1;21(11):1893-1902. doi: 10.5664/jcsm.11800. PMID 40605372

RESULTS

PARTICIPANT FLOW:
Groups:
- Double-Blind Treatment Phase Lower Dose Pitolisant: Stable pitolisant doses of 8.9 mg, 13.35 mg, or 17.8 mg based on age
- Double-Blind Treatment Phase Higher Dose Pitolisant: Stable pitolisant doses of 17.8 mg, 26.7 mg, or 35.6 mg based on age
- Double-Blind Treatment Phase Placebo: Matching placebo tablets
Period: Overall Study
Arm/Group | Double-Blind Treatment Phase Lower Dose Pitolisant | Double-Blind Treatment Phase Higher Dose Pitolisant | Double-Blind Treatment Phase Placebo
Started | 20 | 22 | 23
Completed (Completed Treatment and Completed the DBT Phase) | 18 | 21 | 20
Not Completed | 2 | 1 | 3
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — COVID-19 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-Blind Treatment Phase Lower Dose Pitolisant | Double-Blind Treatment Phase Higher Dose Pitolisant | Double-Blind Treatment Phase Placebo | Total
Number analyzed (Participants) | 20 | 22 | 23 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.1 (5.44) | 13.1 (6.70) | 11.9 (4.31) | 12.4 (5.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 9 | 32
  Male | 9 | 10 | 14 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2 | 4
  Not Hispanic or Latino | 20 | 20 | 21 | 61
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 22 | 23 | 65

OUTCOME MEASURES:

1. Primary Outcome: Excessive Daytime Sleepiness
Description: Change in Epworth Sleepiness Scale for Children and Adolescents (ESS-CHAD) (parent/caregiver version) score from Baseline to Week 11 for pitolisant compared with placebo.
  The score of the ESS-CHAD ranges from 0 to 24. A decrease in score represents an improvement in excessive daytime sleepiness.
Time Frame: Baseline to Week 11
Population: The efficacy population was the modified Intent-to-Treat (mITT) Population, which included all randomized patients who received at least 1 dose of study drug and had both a Baseline assessment and at least 1 post Baseline assessment for a given endpoint analysis during the Double-Blind Treatment Phase.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Double-Blind Treatment Phase Lower Dose Pitolisant | Double-Blind Treatment Phase Higher Dose Pitolisant | Double-Blind Treatment Phase Placebo
Number analyzed (Participants) | 19 | 22 | 21
score on a scale | -3.5 (1.14) | -5.0 (1.07) | -3.9 (1.08)

2. Secondary Outcome: Excessive Daytime Sleepiness
Description: Change in Caregiver Global Impression of Severity for Excessive Daytime Sleepiness.
  The Caregiver Global Impression of Severity for Excessive Daytime Sleepiness is a five-item scale that ranges from "not at all" to "very high likelihood." An assessment of being less likely to fall asleep represents an improvement in the caregiver's overall impression of the patient's excessive daytime sleepiness.
Time Frame: Baseline to Week 11
Reporting Status: Not Posted, anticipated posting 2025-11

3. Secondary Outcome: Clinical Symptoms
Description: Change in Clinical Global Impression of Severity of Overall Clinical Status.
  The Clinical Global Impression of Severity of Overall Clinical Status is a four-item scale that ranges from "normal" to "severely symptomatic." An assessment of less severe symptoms represents an improvement in the clinician's perception of the overall clinical status related to PWS.
Time Frame: Baseline to Week 11
Reporting Status: Not Posted, anticipated posting 2025-11

4. Secondary Outcome: Behavior
Description: Change in Aberrant Behavior Checklist, Second Edition.
  The Aberrant Behavior Checklist-Community, Second Edition, rates 58 specific symptoms on a four-item scale ranging from "not at all a problem" to "the problem is severe in degree." A decrease in score represents an improvement in the caregiver's impression in the patient's problematic behavior.
Time Frame: Baseline to Week 11
Reporting Status: Not Posted, anticipated posting 2025-11

5. Secondary Outcome: Behavioral and Cognitive Rigidity
Description: Change in Montefiore-Einstein Rigidity Scale - Prader-Willi Syndrome (MERS-R-PWS).
  The MERS-R-PWS is a clinician-rated, semi-structured interview conducted with both the patient with PWS and caregiver present. The MERS-R-PWS measures three domains of rigid behavior - behavior, cognitive, and protest. Within each domain, four items are rated on a scale ranging from 0 to 4. A decrease in score represents an improvement in rigid behavior.
Time Frame: Baseline to Week 11
Reporting Status: Not Posted, anticipated posting 2025-11

6. Secondary Outcome: Psychomotor Function
Description: Change in Cogstate Detection Test.
  The Cogstate Detection Test is a computerized test. Accuracy with a faster speed represents an improvement in psychomotor test performance.
Time Frame: Baseline to Week 11
Reporting Status: Not Posted, anticipated posting 2025-11

7. Secondary Outcome: Attention
Description: Change in Cogstate Identification Test.
  The Cogstate Identification Test is a computerized test. Accuracy with a faster speed represents an improvement in attention test performance.
Time Frame: Baseline to Week 11
Reporting Status: Not Posted, anticipated posting 2025-11

8. Secondary Outcome: Working Memory
Description: Change in Cogstate One Back Test.
  The Cogstate One Back Test is a computerized test. Accuracy with a faster speed represents a better working memory test performance.
Time Frame: Baseline to Week 11
Reporting Status: Not Posted, anticipated posting 2025-11

9. Secondary Outcome: Caregiver Burden
Description: Change in 22-Item Zarit Burden Interview.
  The Zarit Burden Interview is a self-reported questionnaire in which caregivers are asked to rate their experience on a five-item scale (0 = "never" and 4 = "nearly always") for 22 questions related to caregiver health and psychological well-being, finances, impact on social life, and relationship with the patient with PWS. A decrease in score represents an improvement in the caregiver's perceived burden.
Time Frame: Baseline to Week 11
Reporting Status: Not Posted, anticipated posting 2025-11

ADVERSE EVENTS:
Time Frame: Data are presented for adverse events occurring after first dose of study drug and up to 30 days after the date of last dose of study drug, for a total of up to 15 weeks.
Description: Data are presented herein for TEAEs. A TEAE is defined as any new adverse event or any worsening of a pre-existing condition that is reported after first dose of study drug and up to 30 days after the date of last dose of study drug.
Arm/Group | Double-Blind Treatment Phase Lower Dose Pitolisant | Double-Blind Treatment Phase Higher Dose Pitolisant | Double-Blind Treatment Phase Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/22 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/22 | 1/23
Other Adverse Events (participants affected / at risk) | 13/20 | 8/22 | 9/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-Blind Treatment Phase Lower Dose Pitolisant (N=20) | Double-Blind Treatment Phase Higher Dose Pitolisant (N=22) | Double-Blind Treatment Phase Placebo (N=23)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind Treatment Phase Lower Dose Pitolisant (N=20) | Double-Blind Treatment Phase Higher Dose Pitolisant (N=22) | Double-Blind Treatment Phase Placebo (N=23)
Anxiety (Psychiatric disorders) | 4 | 1 | 2
Irritability (Psychiatric disorders) | 4 | 1 | 1
Sleep disorder (Psychiatric disorders) | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 2 | 1
COVID-19 (Infections and infestations) | 0 | 3 | 2
Headache (Nervous system disorders) | 3 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0
Hyperphagia (Metabolism and nutrition disorders) | 2 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-08-10): https://cdn.clinicaltrials.gov/large-docs/29/NCT04257929/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-12): https://cdn.clinicaltrials.gov/large-docs/29/NCT04257929/SAP_001.pdf